CLINICAL TRIAL: NCT04185922
Title: Hemopatch to Prevent Lymphatic Leak After Robotic Prostatectomy and Pelvic Lymph Node Dissection: a Randomized Controlled Trial
Brief Title: Hemopatch to Prevent Lymphatic Leak After Robotic Prostatectomy and Pelvic Lymph Node Dissection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Jeremy Yuen Chun TEOH, Assistant Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CRE 2019.419
Record Dates: First submitted 2019-12-03; First posted 2019-12-04 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-06

CONDITIONS: Prostate Cancer
Keywords: Prostate cancer; Hemopatch
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Intervention Model Description: This is a prospective; single-centre phase 3 randomised controlled trial conducted to investigate the efficacy of Hemopatch for preventing lymphatic leak after RARP and BPLND.
Who Masked: Participant
Masking Description: Patients are randomized to receive RARP and BPLND, with or without Hemopatch, with an allocation ratio of 1:1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hemopatch (Experimental): The RARP and BPLND are performed in the usual manner. Towards the end of the operation, Hemopatch is laid over the ends of raw truncated lymphatic tissue.
  Interventions: Device: Hemopatch
- Control (No Intervention): The RARP and BPLND are performed in the usual manner. Hemopatch will not be applied to control group.

INTERVENTIONS:
Device: Hemopatch — As stated in Hemopatch arm description
  Arms: Hemopatch

SUMMARY:
Robotic prostatectomy (RARP) is a surgery for treatment localized prostate cancer. Bilateral pelvic lymph node dissection (BPLND) will also be performed if there is an estimated risk of occult nodal metastases exceeding 5%. BPLND in general is a well-tolerated procedure. Lymphatic leak is one of the possible complications after lymph node dissection (BPLND). Lymphocele is a collection of lymphatic fluid after operation. Hemopatch is a material used during operation that may prevent lymphorrhoea. This is a randomizedcontrolled trial that aims at investigating the application of Hemopatch to raw lymphatic tissue in preventing lymphorrhoea. Patients would be divided into 2 groups: with or without the use of Hemopatch during operation. They will be followed up on day 30 to monitor the course of recovery and any complications.

DETAILED DESCRIPTION:
In prostate cancer patients undergoing robot-assisted radical prostatectomy (RARP), the current European Association of Urology (EAU) prostate cancer guidelines recommend bilateral pelvic lymph node dissection (BPLND) for those with an estimated risk of occult nodal metastases exceeding 5%.(1) In a systematic review of 66 studies involving 275, 269 patients, lymphadenectomy can identify node positive patients who may benefit from adjuvant treatment (2).

BPLND in general is a well-tolerated procedure. However, when complications do occur, significant morbidity results. The benefits of BPLND must be carefully weighed against its potential complications. The most common complication of BPLND is lymphocoele formation. Lymphatic vessels have no muscular layer as opposed to blood vessels. Transection of a blood vessel will lead to vasoconstriction and eventual cessation of bleeding. This is not the case with lymphatic vessels, and transection will lead to prolonged lymphorrhoea. The incidence of lymphocoele varies from series to series, ranging from 0.8% to 33%, depending on the extent of lymphadenectomy, surgical technique, operative approach, and the diagnostic approach (3,4). The most common symptoms are pelvic pain, abdominal distension, lower extremity or scrotal oedema, lower urinary tract symptom, frank bladder outlet obstruction, sepsis and even anastomotic disruption. Prolonged lymphorrhoea lengthens hospital stay, places the patient at risk for nosocomial infection and has significant cost implications for the healthcare system.

Hemopatch is a haemostatic pad consisting of a collagen sheet derived from bovine dermis with an NHS-PEG (pentaerythritol polyethylene glycol ether tetra-succinimidyl glutarate) coated active surface. These two components act together to provide effective tissue adherence, sealing and haemostasis (5). Upon tissue contact, NHS-PEG molecules on the active surface form covalent bonds with tissue proteins. Cross-linking NHS-PEG and proteins forms a hydrogel which acts as an effective tissue seal. Older generation NHS-PEG products in the form of solutions of flowable sealants are quickly washed away by blood or other leaking body fluids, rendering them ineffective in the presence of active bleeding or fluid leakage. Hemopatch is a novel NHSPEG delivery vehicle designed to overcome this limitation. Due to the open pore structure of the collagen, excess tissue fluids are readily absorbed and direct contact of NHS-PEG to tissue surface can be achieved. The collagen pad is optimized to be soft, thin, pliable, and has a high liquid absorption capacity. The pad is resorbed and replaced by host tissue in six to eight weeks with little tissue reaction.

The investigators hypothesise that the application of Hemopatch to raw lymphatic tissue can prevent lymphorrhoea through its unique combination of tissue adherence, sealing and fluid absorption. This can potentially prevent lymphatic leak, reduce drain output and facilitate earlier discharge.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and above
* Able to give informed consent
* Suitable for minimally-invasive surgery

Exclusion Criteria:

* Known allergy or hypersensitivity to any component of Hemopatch®
* Known hypersensitivity to bovine proteins or brilliant blue
* Patients with prior pelvic radiotherapy
* Patients with non-correctable coagulopathy
* Patients who are on anticoagulants
* Contraindication to general anaesthesia
* Previous transurethral resection of the prostate or prostatic surgery
* Untreated active infection

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2020-02-27 (Actual); Primary Completion 2021-07-21 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Total volume of drain output | Three days after the allocated treatment
  Cumulative volume of output from the drain

SECONDARY OUTCOMES:
Operating time | Immediately post-operative
  Duration of operation
Blood loss | Immediately post-operative
  Volume of blood loss during operation
Duration of drainage | Three days after the allocated treatment
  Number of days between insertion and removal of drain
Volume of drainage per post-operative day | Three days after the allocated treatment
  Average volume of drain output per post-operative day
Length of hospital stay | Three days after the allocated treatment
  Patients undergoing robotic radical prostatectomy have an average hospital stay of three days
Transfusion requirement | Three days after the allocated treatment
  Number of units of packed cells being transfused
Lymph node yield | One week after the allocated treatment
  Number of lymph nodes yielded upon pelvic lymph node dissection
30-day complications | Thirty days after the allocated treatment
  Complications which occur within 30 days after the operation

CONTACTS AND LOCATIONS:
Overall Officials: Jeremy Yuen Chun Teoh, MBBS, FRCSEd, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mottet N, Bellmunt J, Bolla M, Briers E, Cumberbatch MG, De Santis M, Fossati N, Gross T, Henry AM, Joniau S, Lam TB, Mason MD, Matveev VB, Moldovan PC, van den Bergh RCN, Van den Broeck T, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Cornford P. EAU-ESTRO-SIOG Guidelines on Prostate Cancer. Part 1: Screening, Diagnosis, and Local Treatment with Curative Intent. Eur Urol. 2017 Apr;71(4):618-629. doi: 10.1016/j.eururo.2016.08.003. Epub 2016 Aug 25. PMID 27568654
- [Background] Fossati N, Willemse PM, Van den Broeck T, van den Bergh RCN, Yuan CY, Briers E, Bellmunt J, Bolla M, Cornford P, De Santis M, MacPepple E, Henry AM, Mason MD, Matveev VB, van der Poel HG, van der Kwast TH, Rouviere O, Schoots IG, Wiegel T, Lam TB, Mottet N, Joniau S. The Benefits and Harms of Different Extents of Lymph Node Dissection During Radical Prostatectomy for Prostate Cancer: A Systematic Review. Eur Urol. 2017 Jul;72(1):84-109. doi: 10.1016/j.eururo.2016.12.003. Epub 2017 Jan 24. PMID 28126351
- [Background] Gilbert DR, Angell J, Abaza R. Evaluation of Absorbable Hemostatic Powder for Prevention of Lymphoceles Following Robotic Prostatectomy With Lymphadenectomy. Urology. 2016 Dec;98:75-80. doi: 10.1016/j.urology.2016.06.071. Epub 2016 Sep 1. PMID 27592524
- [Background] Simonato A, Varca V, Esposito M, Venzano F, Carmignani G. The use of a surgical patch in the prevention of lymphoceles after extraperitoneal pelvic lymphadenectomy for prostate cancer: a randomized prospective pilot study. J Urol. 2009 Nov;182(5):2285-90. doi: 10.1016/j.juro.2009.07.033. Epub 2009 Sep 16. PMID 19762048
- [Background] Lewis KM, Kuntze CE, Gulle H. Control of bleeding in surgical procedures: critical appraisal of HEMOPATCH (Sealing Hemostat). Med Devices (Auckl). 2015 Dec 22;9:1-10. doi: 10.2147/MDER.S90591. eCollection 2016. PMID 26730213